CLINICAL TRIAL: NCT05562583
Title: SAGE-LEAF: Reducing Burden in Alzheimer's Disease Caregivers Through Positive Emotion Regulation and Virtual Support
Acronym: SAGE-LEAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrightOutcome (Industry)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, DerShung Yang, PhD, President, BrightOutcome
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R43AG065080 (NIH)
Record Dates: First submitted 2022-09-18; First posted 2022-10-03 (Actual); Results first posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease and Related Dementias; Caregiver
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (single arm) (Experimental): 5 session self-guided online delivered positive emotion regulation intervention with social components.
  Interventions: Behavioral: SAGE LEAF

INTERVENTIONS:
Behavioral: SAGE LEAF — SAGE LEAF covers 8 skills and each skill has related home-practice activities that "unlock" every week. Each week will consist of 1-2 days of didactic material and 5-6 days of real-life home practice. Participants can access the skills at their own leisure and as often as they'd like within that week. Participants cannot skip modules with didactic material and can only progress to the next lesson if they have completed the current one. However, participants can return to old lessons or exercises if they choose to do so at a later time.

SUMMARY:
The goal of the proposed study, is to adapt a positive emotion intervention for Alzheimer's Disease (AD) caregivers into a self-guided online format that incorporates social connection components and adaptive system feedback mechanisms to promote intervention adherence. Previous tests of the facilitated version of the program, called SAGE-LEAF (Social Augmentation to self-Guided Electronic delivery of the Life Enhancing Activities for Family caregivers), have shown efficacy for improving well-being in dementia caregivers. If effective, the SAGE-LEAF program can be disseminated to Alzheimer's caregivers nationwide through AD treatment and research centers.

DETAILED DESCRIPTION:
The prevalence of Alzheimer's Disease (AD) and other dementias is steadily climbing and predicted to affect as many as 16 million Americans by 2050. In 2016, 59% of dementia caregivers reported experiencing high levels of emotional and physical stress, and the risk that the chronic stress of dementia caregiving places on caregivers for developing a range of physical and mental health issues is extensively documented. Caregiving-related stress contributes to social isolation, loneliness, and physical illness and increases the risk of caregiver death. Interventions for dementia caregivers have primarily focused on reducing negative emotions and burden. However, over the past few decades, it has become clear that positive emotions are uniquely related to better psychological and physical well-being, independent of the effects of negative emotion suggesting that an intervention that specifically targets positive emotion holds promise for improving caregiver well-being and, ultimately, quality of care for the individual living with AD. The investigators' recent randomized trial of the positive emotion skills intervention, delivered by trained facilitators via the web in N = 170 family caregivers of people with dementia resulted in significant improvements in caregiver psychological well being. However, facilitator-delivered interventions are costly and difficult to implement with fidelity on a large scale. Furthermore, a major challenge to advancing behavioral interventions delivered by trained facilitators is assuring fidelity. The investigators have developed a self-guided online version of the intervention that has shown feasibility and acceptability in several samples, but this version does not capture the critical social connection aspects of the facilitator-delivered intervention. The investigators propose to take the next step toward closing the science-to-practice gap for the positive emotion regulation intervention by tailoring the self-guided online version specifically for dementia caregivers that incorporates the social connection components to combat the loneliness and isolation experienced by many Alzheimer's caregivers. The intervention, called SAGE-LEAF (Social Augmentation of self-Guided Electronic delivery of the Life Enhancing Activities for Family caregivers), leverages the lessons learned from the original LEAF project and adapts its positive emotion intervention to AD caregivers in a self-guided format while incorporating social connection components and adaptive system feedback mechanisms to promote intervention adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and over who identify as the primary caregiver of a family member with Alzheimer's Disease
* Co-reside with the family caregiver
* Speak and read English
* Have internet access and a reliable email address

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DerShung Yang, PhD, Principal Investigator — BrightOutcome; Judith T Moskowitz, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Kwok I, Lattie EG, Yang D, Summers A, Grote V, Cotten P, Moskowitz JT. Acceptability and Feasibility of a Socially Enhanced, Self-Guided, Positive Emotion Regulation Intervention for Caregivers of Individuals With Dementia: Pilot Intervention Study. JMIR Aging. 2023 Sep 6;6:e46269. doi: 10.2196/46269. PMID 37672311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a group of individuals who responded to social media advertisements for another caregiver study but were not eligible (3/15, 20%) and from dementia caregiver support groups (12/15, 80%).
Period: Overall Study
Arm/Group | Intervention (Single Arm)
Started | 15
Completed | 10
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Duration of caregiving [Mean (Standard Deviation); unit: years] | 4.27 (2.94)
Diagnosis [Count of Participants; unit: Participants]
  Frontotemporal dementia | 11
  Uncategorized dementia | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Skill Pages in SAGE-LEAF Accessed by a Participant
Description: This is to measure adherence to SAGE-LEAF intervention. Score range: 0-100%. A higher percentage means better adherence to the SAGE-LEAF intervention.
Time Frame: Post-study (week 6)
Measure: Mean (Standard Deviation); unit: Percentage of skill pages
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 15
Percentage of skill pages | 72 (42)

2. Primary Outcome: Willingness to Recommend SAGE-LEAF to Other AD Caregivers
Description: This is to measure the acceptability of SAGE-LEAF. Score range: 1-10. A higher score indicates higher acceptability.
Time Frame: Post-study (week 6)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 8 [6.25 to 9.5]

3. Primary Outcome: System Usability Scale
Description: This is to measure the usability of SAGE-LEAF. Score range: 0-100. A higher score indicates better usability.
Time Frame: Post-study (week 6)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 73.75 [57.5 to 85.63]

4. Secondary Outcome: Zarit Burden Interview
Description: Measuring caregiving burden. Score range: 0-88. Higher scores indicate greater burden.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 15.67 (3.54)

5. Secondary Outcome: Oberst Caregiving Burden Scale - Time
Description: Measuring caregiving burden in terms of time. Score range: 1-5. Higher scores indicate higher levels of caregiver burden.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 3.07 (0.75)

6. Secondary Outcome: Oberst Caregiving Burden Scale - Difficulty
Description: Measuring caregiving burden in terms of difficulty. Score range: 1-5. Higher scores indicate higher levels of caregiver burden.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 2.77 (0.82)

7. Secondary Outcome: Positive Aspects of Caregiving Scale
Description: Measuring positive aspects to caregiving for dementia patients. Score range: 5-45. Higher scores indicate better caregivers' outlook on life and self-affirmations.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 22.23 (9.27)

8. Secondary Outcome: Role Captivity Sub-scale of Caregiver Reaction Assessment
Description: Measuring role captivity in caregiving. Score 1-4. Higher scores indicate stronger feelings of role captivity.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 2.55 (0.7)

9. Secondary Outcome: Overload Sub-scale of Caregiver Reaction Assessment
Description: Measuring the feeling of overload in caregiving. Score 1-4. Higher scores indicate stronger feelings of overload.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 2.65 (0.83)

10. Secondary Outcome: Caregiving Mastery Subscale of the Caregiving Appraisal Measure
Description: Measuring caregiving mastery. Score range: 1-5. Higher scores indicate better caregiving mastery.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 2.66 (0.45)

11. Secondary Outcome: Cohen's Perceived Stress Scale
Description: Measuring perceived stress. Score range: 0-40. Higher scores indicate higher levels of perceived stress
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 7.5 (1.78)

12. Secondary Outcome: Positive Affect in Differential Emotions Scale
Description: Measuring positive emotions. Score range: 1-5. Higher scores indicate higher levels of positive emotions.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 1.82 (0.68)

13. Secondary Outcome: Negative Affect in Differential Emotions Scale
Description: Measuring positive emotions. Score range: 1-5. Higher scores indicate higher levels of negative emotions.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 1.34 (0.72)

14. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Depression
Description: Measuring depression level. Score range: 20-80. Higher scores indicate higher depression levels.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 57.96 (5.05)

15. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Anxiety
Description: Measuring anxiety level. Score range: 20-80. Higher scores indicate higher anxiety levels.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 57.45 (7.96)

16. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Sleep Disturbance
Description: Measuring sleep disturbance level. Score range: 20-80. Higher scores indicate higher levels of sleep disturbance.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 52.73 (7.27)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Meaning and Purpose
Description: Measuring one's sense of life having purpose and that there are good reasons for living. Score range: 20-80. Higher scores indicate hopefulness, optimism, goal-directedness, and feelings that one's life is worthy.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 47.19 (5.63)

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System - Social Isolation
Description: Measuring perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Score range: 20-80. Higher scores indicate higher levels of perception of social isolation.
Time Frame: Pre-study and post-study (week 6)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Single Arm)
Number analyzed (Participants) | 10
score on a scale | 51.27 (5.73)

ADVERSE EVENTS:
Time Frame: The team monitored for adverse events through study completion, i.e., 6 weeks.
Description: Due to the nature and scope of this study, we do not anticipate any adverse events. However, in the case that an adverse event arises, it will be tracked and the PI informed within 24 hours to assess the situation and follow-up. An adverse event form is developed detailing the problem, actions taken, supervisor notes, and follow-up steps performed. The form will be immediately sent to the IRB and NIH. Any action recommended by one of the IRBs will be conveyed to the NIH.
Arm/Group | Intervention (Single Arm)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT05562583/Prot_SAP_000.pdf